CLINICAL TRIAL: NCT00749684
Title: Efficacy and Safety of High-dose Treatment With the Immunomodulator Interferon-α-2b (Intron A®) for the Adjuvant Treatment of Malignant Melanoma.
Brief Title: Efficacy and Safety of High-dose Interferon Alfa-2b (Intron A®) for the Adjuvant Treatment of Malignant Melanoma (Study P04083)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04083
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Results first posted 2011-03-24 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Melanoma
Keywords: interferon-alpha
MeSH Terms: conditions — Melanoma | interventions — Introns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with malignant melanoma at high risk of relapse: Adults with malignant melanoma of the following stages:
  * II and III (>/= 1.5 mm Breslow thickness without distant metastases
  * melanoma with lymph node metastases
  Interventions: Biological: Interferon α-2b

INTERVENTIONS:
Biological: Interferon α-2b — 20 mio IU/m² interferon-α-2b 5x/week intravenously (IV) over the course of 1 month, followed by 10 mio IU/m² interferon-α-2b 3x/week subcutaneously (SC) for 11 months.
  Other Names: Intron A

SUMMARY:
The aim of this observational study is to document the efficacy and tolerability of high-dose interferon therapy in adult participants with malignant melanoma at high risk of relapse and to compare them with the survival times and relapse rates in previous studies (historical control).

DETAILED DESCRIPTION:
Observational study to evaluate the tolerability and efficacy (vs historical controls) of a high-dose therapy scheme with interferon-α-2b (IntronA®):

Adjuvant treatment with interferon-α-2 has been demonstrated in a number of studies to have an antiproliferative effect on malignant melanoma. In these cases a response rate of up to 20% could be achieved with a dose of 10 million IU or more 3x/week or daily. Kirkwood et al. showed in a study carried out in ECOG (the Eastern Cooperative Oncology Group, study no. 1684) that there was a clear and significant survival advantage versus the observation group with the following dose:

20 mio IU/m² interferon-α-2b (IntronA®) 5x/week iv over the course of one month followed by 11 months with 10 mio IU/m² 3x/week sc.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants
* Age 18-70 years
* Malignant melanoma stage II or III (>/= 1.5 mm tumor thickness, no distant metastases or Malignant melanoma with lymph node metastases or Lymph node metastases with unknown primary tumor
* An excision border of at least 2 cm around the primary tumor
* Therapy must start within 12 weeks after surgery of the tumor/of the lymph node metastases
* ECOG status 0-1 (= Karnofsky Index >/= 80)
* Laboratory parameters

  * Hematocrit >= 33%
  * Leukocytes >= 3000/μl
  * Thrombocytes >= 100000/μl
  * Alanine aminotransferase(ALT) <= 2x normal values
  * Bilirubin <= 2x normal values

Exclusion Criteria:

* Known allergy to one of the medications or any of its component parts
* Refusal on the part of participants capable of childbearing to use a reliable contraceptive
* Lactating mothers
* Presence of distant metastases
* Another primary tumor of different histological origin than corresponding to the indication (except when the relapse-free interval is > 5 years, or the tumor is a cervical carcinoma in situ, a basal cell carcinoma or cutaneous squamous cell carcinoma)
* Participants on corticosteroid treatment or treatment with an immunomodulating substance
* Preexisting psychiatric illness, particularly serious depression
* Prior adjuvant radio-, chemo-, or immuno-therapy
* Treatment with an investigational drug within the prior 30 days
* Participant history that includes cardiac arrhythmia, cardiac insufficiency requiring treatment, or anthracycline administration
* Myocardial infarction within the prior year
* An unstable medical condition (apart from the indication) that in the judgment of the investigating physician excludes the participants from the study
* Psoriasis (a relative exclusion criterion, since interferon can aggravate psoriasis; decision to be based on risk/benefit analysis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants in Austria with malignant melanoma at high risk of relapse
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 1996-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female participants, with malignant melanoma Stage II or III (>1.5 mm tumor thickness, no distant metastasis) or malignant melanoma with evidence of lymph node metastis or lymph node metastasis of malignant melanoma at unknown primary tumor, primary tumor has to be surgically resected within 2 months after first biopsy/excision.
Period: Overall Study
Arm/Group | Adults With Malignant Melanoma at High Risk of Relapse
Started | 138
Completed | 56
Not Completed | 82
Not completed — Death | 1
Not completed — Adverse Event | 27
Not completed — Participant's Wish | 10
Not completed — Not Documented | 1
Not completed — Progressive Desease | 31
Not completed — Therapy according to protocol + AE | 2
Not completed — AE+discontinuation on participants wish | 1
Not completed — Missing | 9

BASELINE CHARACTERISTICS:
Arm/Group | Adults With Malignant Melanoma at High Risk of Relapse
Number analyzed (Participants) | 138
Age, Continuous [Median (Standard Deviation); unit: participants]
  Total | 48.83 (12.72)
  Male | 49.15 (12.91)
  Female | 48.27 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 (12.49)
  Male | 88 (12.91)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Recurrence
Description: Number of participants with disease recurrence was being measured.
Time Frame: Throughout 12 months of treatment and 24 months of follow-up
Population: 138 participants with malignant melanoma, 88 male participants and 50 female participants were evaluated.
Measure: Number; unit: participants
Arm/Group | Adults With Malignant Melanoma at High Risk of Relapse
Number analyzed (Participants) | 138
participants | 52

2. Primary Outcome: Relapse Free Survival Time
Description: Median time to recurrence according to Kaplan Maier evaluation
Time Frame: Throughout 12 months of treatment and 24 months of follow-up
Measure: Median (Full Range); unit: months
Arm/Group | Adults With Malignant Melanoma at High Risk of Relapse
Number analyzed (Participants) | 138
months | 54.1 [0 to 60]

ADVERSE EVENTS:
Arm/Group | Interferon Alfa-2b
Serious Adverse Events (participants affected / at risk) | 11/138
Other Adverse Events (participants affected / at risk) | 75/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Alfa-2b (N=138)
DEATH (General disorders) | 1 (1)
SARCOIDOSIS (Immune system disorders) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1)
EPILEPSY (Nervous system disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 2 (2)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
VENOUS THROMBOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Alfa-2b (N=138)
LEUKOPENIA (Blood and lymphatic system disorders) | 13 (20)
NAUSEA (Gastrointestinal disorders) | 12 (13)
FATIGUE (General disorders) | 13 (20)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 12 (17)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 17 (19)
TRANSAMINASES INCREASED (Investigations) | 8 (9)
DECREASED APPETITE (Metabolism and nutrition disorders) | 7 (9)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 7 (7)
HEADACHE (Nervous system disorders) | 9 (9)
DEPRESSION (Psychiatric disorders) | 14 (14)
ALOPECIA EFFLUVIUM (Skin and subcutaneous tissue disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No